CLINICAL TRIAL: NCT06755203
Title: Evaluating the Impact of Operating Room Simulations on Communication Skills and Patient Safety
Brief Title: Evaluating the Impact of Operating Room Simulations on Communication Skills and Patient Safety (EIORS-CPS)
Acronym: EIORS-CPS
Status: Recruiting | Type: Observational
Sponsor: King Saud Medical City (Other Government)
Responsible Party: Principal Investigator, Walid Mohamed Ragab Mohamed Badwi, A resident in anesthesia department, king Saud Medical City Teacher and Instructor in (Basic Anesthesia and Resuscitation-MEDI 045) King Saud University College of Medicine / anesthesia department Undergraduate Education Organizer, King Saud Medical City
Other Study IDs: King Saud Medical City; IRB Ref. No. 24/1145/IRB (Other: College of Medicine, KSU, Riyadh, Saudi Arabia)
Record Dates: First submitted 2024-12-16; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Patient-Centered Care; Competency-Based Education
Keywords: Patient safety; WHO Surgical Safety Checklist; Team communication; Stress management; Protocol adherence; Risk assessment; Operating room simulations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Simulation Training Group: Participants will engage in operating room simulations designed to improve communication skills, stress management, and adherence to the WHO Surgical Safety Checklist.
  Interventions: Other: Operating Room Simulation Training

INTERVENTIONS:
Other: Operating Room Simulation Training — The intervention involves high-fidelity OR simulations focusing on critical areas of patient safety, including:
  Communication Skills: Emphasizing clear communication during surgical procedures.
  Stress Management: Training participants to manage stress effectively in high-pressure situations.
  Protocol Adherence: Practicing adherence to the WHO Surgical Safety Checklist. Risk Assessment: Identifying and mitigating potential safety risks in simulated scenarios
  Other Names: Patient Safety Simulation

SUMMARY:
Simulation-based training has emerged as a valuable tool for enhancing communication skills among healthcare professionals. This study aimed to evaluate the impact of operating room (OR) simulations on the development of communication skills for patient safety. The study focused on two key areas: the development of communication skills for patient-centered care and the role of the WHO Surgical Safety Checklist in enhancing communication and patient safety during simulations.

DETAILED DESCRIPTION:
This study will provide valuable insights into student preferences for logbook formats in anesthesiology education, specifically within the MEDI 045 course. By comparing Excel sheet logbooks with traditional paper logbooks, it aims to elucidate how different documentation methods impact student engagement, satisfaction, and learning outcomes.

Understanding these preferences is crucial, as logbooks are not merely administrative tools but integral components of the educational experience that promote reflection, accountability, and skill development in clinical practice.

The findings will contribute to existing knowledge by identifying specific advantages and disadvantages of each format, highlighting the aspects that enhance or hinder student learning. Moreover, the research will inform curriculum designers and educators about effective strategies for logbook implementation, ultimately leading to improved educational tools that better align with students' needs

ELIGIBILITY:
Inclusion Criteria:

Participants must be medical students enrolled in the MEDI 045 course at King Saud University.

Must have prior exposure to basic patient safety and communication skills training.

Age: 18-25 years. Students must voluntarily consent to participate in the study and complete the required simulations and assessments.

Exclusion Criteria:

Students who have already completed formal simulation-based training on communication or patient safety outside the MEDI 045 curriculum.

Students are unable to participate in simulation sessions due to scheduling conflicts or medical reasons.

Participants were unwilling to provide informed consent.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population includes medical students enrolled in the MEDI 045 course at King Saud University. These students are actively engaged in clinical education and exposed to scenarios requiring the development of communication skills and adherence to the WHO Surgical Safety Checklist.
  Key Characteristics:
  Academic Level: Medical students introduced to clinical practices in anesthesia.
  Training Context: Students participating in structured educational activities, such as logbook maintenance and simulation-based learning.
  Sample Size: Approximately 109 students to ensure robust analysis of communication skills and logbook preferences.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Estimated)
Dates: Start 2024-03-03 (Actual); Primary Completion 2025-01-25 (Estimated); Study Completion 2025-02-25 (Estimated)

PRIMARY OUTCOMES:
Improving Patient Safety Training through Simulation | 7-8 months
  Evaluate the effectiveness of simulation-based training in promoting patient safety with a focus on:
  Authenticity: Scenarios mirroring real operating room environments. Stress Management & Communication: Improving interpersonal dynamics, team synergy, and decision-making under pressure.
  Protocol Compliance & Risk Evaluation: Ensuring adherence to patient safety best practices.
  WHO Surgical Safety Checklist: Enhancing communication and protocol adherence. Evaluation Tool: Patient Safety Simulation Assessment Scale (PSSAS).
  Scale Range: 0-10
  Criteria:
  0-3: Minimal improvement. 4-6: Moderate improvement. 7-8: Significant improvement. 9-10: Excellent improvement. Higher scores indicate better outcomes.

SECONDARY OUTCOMES:
Improvement in Communication Skills during Simulations | 7-8 months
  Evaluate the enhancement of communicative competencies, placing particular emphasis on:
  Clarity of Communication: The proficiency in transmitting information with efficacy. Teamwork: The synergy and coordination exhibited within the group. Adherence to Structured Communication Protocols: The implementation of standardized tools such as SBAR (Situation-Background-Assessment-Recommendation). Measurement Tool: A bespoke Structured Communication Skills Evaluation Checklist (SCSEC) will be employed. Scale Range: 0-10 Scoring Criteria: 0-3: Insignificant clarity and teamwork, accompanied by inadequate adherence to protocols. 4-6: Moderate clarity and teamwork, coupled with partial compliance to protocols. 7-8: Robust clarity and teamwork, characterized by commendable adherence to protocols. 9-10: Exemplary clarity and teamwork, demonstrating complete adherence to protocols. Elevated scores signify superior outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- King Saud University , College of Medicine, Anesthesia Department, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
At this time, there are no plans to share individual participant data (IPD) publicly. The study will retain data within the institution for research purposes only.